CLINICAL TRIAL: NCT02032849
Title: Air-impingement Manipulation to Clear Subglottic Secretion Compared With Drainage Tube in Prolonged Intubated Patients, a Randomized Controlled Trial.
Brief Title: Air-impingement Manipulation to Clear Subglottic Secretion Compared With Drainage Tube in Prolonged Intubated Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Jie Li, RRT-NPS, Beijing Chao Yang Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: BJCYHRT-001
Record Dates: First submitted 2013-12-30; First posted 2014-01-10 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-08

CONDITIONS: Ventilator Associated Pneumonia
Keywords: ventilator associated pneumonia; subglottic secretion drainage; manual air-impingement operation; prolonged intubation
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- subglottic secretion drainage (Active Comparator): The conventional method with a special tube to drainage subglottic secretion
  Interventions: Procedure: Manual air-impingement operation
- Manual air-impingement operation (Experimental): A method which we invented to clear subglottic secretion
  Interventions: Device: subglottic secretion drainage

INTERVENTIONS:
Procedure: Manual air-impingement operation — A method which we invented to clear subglottic secretion
  Arms: subglottic secretion drainage
Device: subglottic secretion drainage — The conventional method with a special tube to drainage subglottic secretion
  Arms: Manual air-impingement operation

SUMMARY:
This is a randomized controlled trial compared two methods to drainage subglottic secretion in prolonged intubated patients.After enrolled, patients are randomized assigned to intermittent subglottic secretion drainage group and air-impingement manipulation group.

DETAILED DESCRIPTION:
Ventilator-associated pneumonia (VAP) is the most frequent infection occurring in patients who are admitted to the ICU. The accumulation of respiratory secretions in the subglottic space is a well-proven cause of VAP. Therefore, prevention should include the aspiration of secretions from the subglottic space. Investigators invented a manual method with high-flow air produced by resuscitator to impinge secretion from the subglottic space to oral cavity. This method has been granted as a patent by Chinese national intellectual property patent office, it has been used in investigators' daily work for more than 10 years and more than 20 Chinese ICUs have used it everyday. Investigators want to compare it with conventional method which uses a special intubation tube with an independent dorsal lumen to suction subglottic secretion.

ELIGIBILITY:
Inclusion Criteria:

Should meet all the criteria:

1. Intubation less than 24 hours before admitting respiratory intensive care unit;
2. Anticipated intubation for more than 72 hours;
3. Anticipated survival time is more than 2 weeks

Exclusion Criteria:

Meet any of these criteria:

1. PEEP≥10cmH2O or FiO2≥0.8;
2. unstable hemodynamics;
3. severe bulla and pneumothorax;
4. enrolled in other study;
5. cuff leak test is positive.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2014-02; Primary Completion 2016-06 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with ventilator-associated pneumonia | Up to 28 days

SECONDARY OUTCOMES:
ICU mortality | Participants will be followed for the duration of ICU stay, an expected average of 4 weeks

OTHER OUTCOMES:
Invasive ventilation duration | Participants will be followed for the duration of invasive ventilation, an expected average of 7-10 days

CONTACTS AND LOCATIONS:
Overall Officials: Jie Li, Master, Principal Investigator — Beijing Chao Yang Hospital
Locations (1):
- Beijing Chaoyang hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Li Y, Yuan X, Sun B, Li HC, Chu HW, Wang L, Zhao Y, Tang X, Wang R, Li XY, Tong ZH, Wang C. Rapid-flow expulsion maneuver in subglottic secretion clearance to prevent ventilator-associated pneumonia: a randomized controlled study. Ann Intensive Care. 2021 Jun 24;11(1):98. doi: 10.1186/s13613-021-00887-5. PMID 34165661